CLINICAL TRIAL: NCT03430726
Title: The ProbGut Study: Effects of Probiotics on the Gut Microbiota of Healthy Children
Brief Title: ProbGut: Probiotics on the Healthy Gut Microbiota
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Kim Chau, Principal Investigator, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROBGUT
Record Dates: First submitted 2018-01-25; First posted 2018-02-13 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Probiotics; paediatrics; gut microbiota

STUDY DESIGN:
Intervention Model Description: All eligible participants will be assigned to receive the commercially available yogurt drink containing a multi-strain probiotic, Bio-Kidz® (12.5 billion CFU/98g; Lactobacillus acidophilus CL1285®, Lactobacillus casei LBC80R® and Lactobacillus rhamnosus CLR2®), daily for 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Kids Probiotic Yogurt Drink Group (Experimental): Healthy children will be given a commercially available yogurt drink containing a multi-strain probiotic, Bio-Kidz® (12.5 billion CFU/98g; Lactobacillus acidophilus CL1285®, Lactobacillus casei LBC80R® and Lactobacillus rhamnosus CLR2®), daily for 14 days.
  Interventions: Other: Probiotic yogurt drink

INTERVENTIONS:
Other: Probiotic yogurt drink — Food product; yogurt drink containing a multi-strain probiotic.
  Other Names: Bio-Kidz® (12.5 billion CFU/98g; Lactobacillus acidophilus CL1285®, Lactobacillus casei LBC80R® and Lactobacillus rhamnosus CLR2®)

SUMMARY:
In adults, probiotics have been shown to have no effect on the microbial composition and the beneficial effects are only transient. However, the gut microbiota of young children is less stable and more impressionable. The aim of this study is to examine the effects of probiotics on the developing microbiota in early life and to determine whether a young child's microbiota may be less resilient to probiotic-induced changes and possibly resulting in longer lasting probiotic effects compared to adults.

DETAILED DESCRIPTION:
Probiotics are live microorganisms that have been associated with health benefits. However, probiotic effects have not been shown to persist beyond discontinuation of use in adults. The intake of probiotics during the critical window of gut microbiota development in young children, however, may allow for a longer duration of persistence of probiotic bacteria and more stable changes in microbial composition possibly resulting in stable engraftment of the probiotic strains. This study aims is to examine the effect of a 14-day course of a commercially available probiotic yogurt drink on the composition, diversity, and changes in immune biomarkers (e.g. human beta-defensin-2 and calprotectin) of the gut microbiota of healthy children. As well, to assess whether the probiotic strains persists after discontinuation of intake and whether engraftment occurs. By understanding the impact of probiotics on the gut microbiota, we will better understand the mechanism by which probiotics exert their beneficial effects. This may help guide probiotic selection based on the potential short- and long-term effects on the commensal microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be healthy children between 1 to 3 years of age.

   * Participants will be considered healthy on entry into the study if they did not have a history of chronic gastrointestinal issues, including chronic or frequent episodes of diarrhea (>3 bowel movements/day for 3 consecutive days) during the month prior to enrolment.
2. Mother of participant is able to communicate in English (read, write, speak), as she will be required to provide her personal and medical history.

Exclusion Criteria:

1. Lactose or milk protein intolerance, or strawberry anaphylaxis, or allergies to dried citrus pulp, or any other components of the study product.
2. Immuno-compromised children (e.g. heart or kidney transplant, complex care, sickle cell disease) or those on immunosuppressive agents (e.g. chemotherapy agents, oral prednisone).
3. Children with known or potentially compromised gut integrity (e.g. short gut, Inflammatory Bowel Disease, Celiac, nasogastric, naso-jejunal or gastrostomy tube).
4. Children admitted to a medical or surgical subspecialty unit.
5. Children on antimicrobial therapy within 30 days prior to enrolment.
6. Children on an alternative probiotic within 30 days prior to enrolment.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Composition and Diversity of Gut Microbiota | Baseline, 30 days and 90 days
  Change in microbial community (e.g. alpha and/or beta diversity) post-probiotic
Levels of Fecal Biomarkers - beta-defensins-2 (hBD-2) | Baseline, 21 days, 30 days, and 90 days
  Change in levels of beta-defensins-2 (hBD-2)
Levels of Fecal Biomarkers - Fecal Calprotectin | Baseline, 21 days, 30 days, and 90 days
  Change in levels of Fecal Calprotectin

SECONDARY OUTCOMES:
Duration of Persistence (DOP) | 90 days post intervention
  Measure detectable levels of probiotic strains post-treatment
Occurrence of Adverse Events | Through study completion, an average of 121 days.
  Measure the occurrence and description of adverse events associated with probiotic use

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No